CLINICAL TRIAL: NCT00534729
Title: Organ Preservation: Weekly Carboplatin & Taxol w/Concurrent RT for Locally Advanced Laryngeal & Hypopharyngeal CA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC#0971-024
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2016-01

CONDITIONS: Laryngeal Neoplasms; Hypopharyngeal Neoplasms
Keywords: Organ Preservation; Carboplatin; Taxol; RT; laryngeal & Hypopharyngeal CA; Locally advanced laryngeal & Hypopharyngeal CA
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Weekly Carboplatin & Taxol w/concurrent RT — Chemotherapy

SUMMARY:
Organ Preservation: Weekly Carboplatin & Taxol w/concurrent RT for locally advanced laryngeal & Hypopharyngeal CA

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced laryngeal & Hypopharyngeal CA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
safety | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Al-Rajhi, MD, Principal Investigator — KFSH&RC
Locations (1):
- KFSH&RC, Riyadh, Saudi Arabia